CLINICAL TRIAL: NCT00412230
Title: The Role of Insulin Resistance in Gestational Hypertension and in Preeclampsia.
Brief Title: Insulin Resistance and Hypertensive Disorders in Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Messina (Other)
Responsible Party: Rosario D'Anna, University of Messina
Other Study IDs: 120254
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Hypertension in Pregnancy; Diabetes Mellitus in Pregnancy
Keywords: Pre-eclampsia; Gestational diabetes; Insulin resistance; hypertension in pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Diabetes, Gestational; Pre-Eclampsia; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- no treatment
- 2

SUMMARY:
The purpose of this study is to determine whether insulin resistance might affect the pathogenesis of hypertensive disorders in pregnancy since midtrimester. Furthermore, markers of vascular and placental injuries, of oxidative stress and inflammation will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* PCOS, BMI>/=30
* previous pregnancy affected by hypertension or gestational diabetes
* thrombophilia
* Type I or II diabetes mellitus
* autoimmune diseases
* twin pregnancy
* renal diseases
* previous pre-eclampsia in relatives

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant outpatients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2006-10; Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosario D'Anna, Associate Professor, Principal Investigator — University of Messina
Locations (1):
- University Hospital, Messina, Italy